CLINICAL TRIAL: NCT06422312
Title: Clinical Investigation to Evaluate the Effectiveness of the Redpine Disposable Scope Compared to Standard Reusable Scope for Flexible Cystoscopy.
Brief Title: A Study Comparing a Disposable Flexible Cystoscope With Reusable Scopes in Adult Patients.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: A change in marketing strategy resulted in a decision to not complete the trial.
Sponsor: Guangzhou Red Pine Medical Instrument Co., Ltd. (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other); University of Washington (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Yair Lotan, MD, Professor Vice Chair of Clinical Affairs Chief of Urologic Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USA001
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer; Bladder Stone; Bladder Outlet Obstruction; Renal Stone; Renal Disease
Keywords: cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder Calculi; Urinary Bladder Neck Obstruction; Nephrolithiasis; Kidney Diseases | interventions — Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Participants in this arm will receive cystoscopy using the clinic's standard of care flexible reusable cystoscope of the urologist's choice.
  Interventions: Device: Cystoscopy with standard of care flexible reusable scope
- Intervention (Experimental): Participants in this arm will receive cystoscopy using the Redpine® Rflex endoTMHD Cysto scope.
  Interventions: Device: Cystoscopy with RedPine flexible disposable cystoscope

INTERVENTIONS:
Device: Cystoscopy with RedPine flexible disposable cystoscope — Use of a disposable flexible cystoscope to visualize the urethra and bladder, take biopsies, and remove stents.
  Arms: Intervention
Device: Cystoscopy with standard of care flexible reusable scope — Use of a reusable flexible cystoscope to visualize the urethra and bladder, take biopsies, and remove stents
  Arms: Control

SUMMARY:
This study will compare the time required for a cystoscopy procedure in adult participants using the Redpine® Rflex endo(trademark) High-Definition Cystoscope or the site's standard of care reusable flexible cystoscope in participants requiring urethral stent removal.

DETAILED DESCRIPTION:
This randomized study will compare the cumulative procedure time between cystoscopy performed with the Redpine® Rflex endo(trademark) High-Definition Cystoscope and the site's standard of care reusable flexible cystoscope in adult study participants requiring cystoscopy for visualization of and/or intervention on the urinary bladder. The study will evaluate the user experience and product performance during cystoscopic procedures. Participant experience, tolerance to the procedure, and any differences in adverse events between disposable and reusable scope will be evaluated. The hypothesis is that the RedPine cystoscope will perform as well as reusable scopes and will have a shorter cumulative procedure time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 18 years old
2. Patient undergoing routine flexible cystoscopy
3. No active urinary tract infection
4. Subject is willing and able to sign informed consent and HIPAA authorization.

Exclusion Criteria:

1. Known unpassable urethral stricture
2. Febrile patient with active urinary tract infection (UTI)
3. Subjects with acute infection (acute urethritis, acute prostatitis, acute epididymitis)
4. Subject with severe coagulopathy
5. Subject is pregnant or female with reproductive capability who is unwilling to have a pre-procedure pregnancy test and use birth control.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative Procedure Time | 30 minutes
  To compare the Cumulative Procedure Time between cystoscopy performed with the Redpine® Rflex endo(trademark) High Definition (endoTMHD) Cysto scope and the site's Standard of Care reusable flexible cystoscope as measured by:
  * Scope preparation for procedure
  * Actual procedure time (insertion of cystoscope to complete bladder examination) and
  * Time to dispose of or prepare for reprocessing of cystoscopy equipment.

SECONDARY OUTCOMES:
User experience and product performance during cystoscopic procedures | within 24 hours
  Physician satisfaction, rated on a five-point scale.
  Scale Name Very Difficult Very Easy Outcome
  Ease of insertion 1 5 5 = Better
  Ability to visualize anatomical landmarks and/or urothelium changes 1 5 5 = Better
  Perception of image quality 1 5 5 = Better
  Maneuverability in the bladder 1 5 5 = Better
  Overall Acceptability Yes/No
Participant comfort during the procedure | 30 minutes
  Participants will be interviewed using a questionnaire. Pain Intensity Please respond to the question by marking one box.
  How would you rate your pain on average? 0 1 2 3 4 5 6 7 8 9 10 No pain Worst imaginable pain
RedPine Cystoscope Conversion Rate | 30 minutes
  Rate of conversion to a reusable cystoscope for those subjects randomized to the REDPINE cystoscope.
Device Failure Rate | 30 minutes
  Device failure leading to a serious adverse event (SAE), termination of the procedure, or conversion to a reusable cystoscope.

OTHER OUTCOMES:
Safety Endpoints | 4 to 10 days
  Safety will be assessed based on the incidence rates of adverse events based on the seriousness and relatedness to the device and/or procedure.
  1) All urologic adverse events, both device and procedure related, during the cystoscopy procedure through 7 (+/- 3) days post-procedure.
  The subject will be asked if they have had:
  1. any signs or symptoms of a UTI
  2. any untoward effects post-procedure, including by not limited to
     1. gross hematuria last longer than 3 days post-procedure
     2. pain with urination lasting longer than 3 days post-procedure
     3. cloudy urine noted greater than one day post-procedure
     4. fever/chills or a diagnosis of UTI or other illness within the time since the cystoscopic procedure.
        2) All reported device and/or procedural related adverse events through 7 (+/- 3) days post- procedure 3) All Serious Adverse Events (SAEs) through 7 (+/- 3) days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - Pennsylvania State University, Hersey, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samplaski MK, Jones JS. Two centuries of cystoscopy: the development of imaging, instrumentation and synergistic technologies. BJU Int. 2009 Jan;103(2):154-8. doi: 10.1111/j.1464-410X.2008.08244.x. Epub 2008 Dec 8. PMID 19076146
- [Background] O'Sullivan DC, Chilton CP. Flexible cystoscopy. Br J Hosp Med. 1994 Apr 6-19;51(7):340-5. PMID 8081563
- [Background] Poulton LJ, Joyce AD. Flexible cystoscopy: Training and Assessment Guideline. Br Assoc Urol Nurses. 2012;(November).
- [Background] Pillai PL, Sooriakumaran P. Flexible cystoscopy: a revolution in urological practice. Br J Hosp Med (Lond). 2009 Oct;70(10):583-5. doi: 10.12968/hmed.2009.70.10.44626. PMID 19966704
- [Background] Kadi N, Menezes P. ABC of flexible cystoscopy for junior trainee and general practitioner. Int J Gen Med. 2011;4:593-6. doi: 10.2147/IJGM.S20267. Epub 2011 Aug 19. PMID 21887113
- [Background] Steinberg. Cystoscopy in Bladder Carcinoma [Internet]. Medscape. 2015 [cited 2018 Jan 18]. Available from: https://emedicine.medscape.com/article/1950345-overview
- [Background] Doizi S, Kamphuis G, Giusti G, Palmero JL, Patterson JM, Proietti S, Straub M, de la Rosette J, Traxer O. First clinical evaluation of a new single-use flexible cystoscope dedicated to double-J stent removal (Isiris): a European prospective multicenter study. World J Urol. 2017 Aug;35(8):1269-1275. doi: 10.1007/s00345-016-1986-0. Epub 2016 Dec 17. PMID 27988848